CLINICAL TRIAL: NCT02764827
Title: Comparison of Skin Prick Testing Results of Local and Imported Pollen Allergen Extracts (Bermuda ,Johnson Grasses and Careless Weed) With Specific IgE Levels.
Brief Title: Comparison of Skin Prick Testing Results of Local and Imported Pollen Allergen Extracts and Specific IgE
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: Si246/2556
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Immediate Type Hypersensitivity
Keywords: skin prick test; grass and weed pollens

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Pollen sensitization — Skin prick test with local and imported Bermuda, Johnson and careless weed allergen extracts at concentration of 10,000, 3,000, 1,000 and 300 AU/mL and measure specific IgE levels

SUMMARY:
Pollen allergen extracts are prepared locally and checked for efficacy by comparison to imported allergens and specific IgE.

DETAILED DESCRIPTION:
Skin prick test (SPT) and specific IgE (sIgE) are approved for evaluation of allergen sensitization. Local allergen extracts are cheaper and more available but need standardization. Pollen allergen extracts: Bermuda, Johnson and careless weed are locally prepared and compared mean wheal diameter of skin prick test to imported allergens and also to specific IgE.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to Bermuda or Johnson or careless weed

Exclusion Criteria:

* Chronic diseases such as heart disease, liver, renal and severe sepsis
* Severe allergic symptoms such as anaphylaxis
* Extensive skin rashes
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People 18-60 years of age who recently have positive skin prick test to grass pollen or careless weed are pricked with local and imported Bermuda grass, Johnson grass and careless weed allergen extracts. Specific IgE levels are also measured at the same day.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean wheal diameter of local and imported grass and weed pollens | 18 months
  compare mean wheal diameter of skin prick test of different concentration among local, imported allergen extract and specific IgE levels of Bermuda grass, Johnson grass and careless weed
sIgE levels of Bermuda grass,Johnson grass and careless weed | 18 months
  Measure level of sIgE of Bermuda grass,Johnson grass and careless weed and compare to SPT results

IPD SHARING:
Plan to Share IPD: No